CLINICAL TRIAL: NCT03148951
Title: Effect of Neutrophil /Lymphocyte Ratio (NLR) and Mean Platelet Volume (MPV) on Early Postoperative Outcome in Lower Extremity Arthroplasty Operations
Brief Title: Effect of NLR and MPV on Early Postoperative Outcome in Lower Extremity Arthroplasty Operations
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, İlker Onguc Aycan, Associated Professor, Akdeniz University
Other Study IDs: MANLOP
Record Dates: First submitted 2017-05-02; First posted 2017-05-11 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Knee Arthropathy
Keywords: MPV; NLR; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Group 1: patients receiving general anesthesia and having a postoperative pain VAS score equal to or below 50 at 1st, 6th, 12th nd 24th hours the pain sores will be evaluated at 4 time intervals and so the number of patients in every group may change at every time interval.
- Group 2: Group 2: patients receiving general anesthesia and having a postoperative pain VAS score equal to or above 60 at 1st, 6th, 12th nd 24th hours the pain sores will be evaluated at 4 time intervals and so the number of patients in every group may change at every time interval.
- Group 3: Group 3: patients receiving regional (spinal) anesthesia and having a postoperative pain VAS score equal to or below 50 at 1st, 6th, 12th nd 24th hours the pain sores will be evaluated at 4 time intervals and so the number of patients in every group may change at every time interval.
- Group 4: Group 4: patients receiving spinal anesthesia and having a postoperative pain VAS score equal to or above 60 at 1st, 6th, 12th nd 24th hours the pain sores will be evaluated at 4 time intervals and so the number of patients in every group may change at every time interval.

SUMMARY:
In the planned study the investigators want to evaluate the relation between postoperative complications and minor/ major morbidities, mortality and Mean Platelet Volume (MPV) and Neutrophil/ lymphocyte (N/L) ratio.

DETAILED DESCRIPTION:
* In this study the investigators aim to determine the relation between the MPV and N/L ratio and the incidence of postoperative adverse events and complications in patients undergoing knee arthroplasty.
* In this study only the laboratory tests that are routinely used for the operative patients are going to be used and no extra tests will be performed. The study will begin after the postoperative blood samples are collected for routine laboratory measurements. The patients will be allocated to 4 groups according to the type of anesthesia and VAS scores. Preoperative and postoperative peripheral blood total whole blood MPV and N/L ratio and 1st 6th 12th ve 24th hours VAS scores and complications, morbidities and mortality will be recorded. The patients will receive analgesics according to the routine practice in the ward and the doses of analgesics given will be recorded at 1st 6th 12th ve 24the hours wil be recorded.
* Statistical analysis: the numerical variables will be analyzed tested with Kolmogorov-Smirnov test for normality. For the parametric variables that are normally distributed t-test will be used for the comparison between groups. For the parametric variables that are not normally distributed Mann Whitney-U test will be used. All the categorical variables will be evaluated with q- square tests. A p value < 0.05 will be determined as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* knee arthroplasty patients with general or spinal anesthesia.

Exclusion Criteria:

* patients not giving consent
* reoperations
* patients having inflammatory disease
* infection in the knee
* sepsis
* bleeding disorders
* hematologic diseases,
* using steroids.
* trauma
* fracture patients,
* bilateral knee prothesis
* combined surgery procedures
* patients needing perioperative transfusions
* uncooperative patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients undergoing knee arthroplasty in 3 years period with general or spinal anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 754 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
postoperative VAS (visual analogue scale) score | VAS score at postoperative twenty-forth hours will be evaluated
  postoperative visual analog scale score for pain evaluation 0,10,20,30,40,50,60,70,80,90,100)

SECONDARY OUTCOMES:
analgesic drugs | total dose of analgesic drugs required at twenty four hours will be evaluated
  analgesic drugs given according to the routine practice in the ward
postoperative major morbidities | at postoperative first, sixth, twelfth and twenty-forth hours
  postoperative Myocardial Infarction (MI), Acute Kidney Injury(AKI), and Cerebrovascular Events (CVO)s.

OTHER OUTCOMES:
postoperative side effects | at postoperative first, sixth, twelfth and twenty-forth hours
  nausea, vomiting, abdominal pain, agitation, head ache, muscular weakness, dizziness,hiccups, bronchospasm, bradycardia, itching, urinary retention,

CONTACTS AND LOCATIONS:
Overall Officials: Ilker o Aycan, asso prof, Principal Investigator — Akdeniz University Hospital
Locations (1):
- AkdenizU, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The role of mean platelet volume in patients with non-specific abdominal pain in an emergency department — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4607690/pdf/PG-10-24573.pdf
- See also: Neutrophil/Lymphocyte Ratio as a Predictor of In-Hospital Major Adverse Cardiac Events, New-Onset Atrial Fibrillation, and No-Reflow Phenomenon in Patients with ST Elevation Myocardial Infarction — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4750894/pdf/cmc-10-2016-019.pdf